CLINICAL TRIAL: NCT01117090
Title: Feasibility of Measuring Cerebrospinal Fluid (CSF) Signatures in Subjects With Intrathecal Catheter-Related Problems
Brief Title: Measuring Signatures in the Fluid Surrounding the Spinal Cord in Patients Who Have Problems With Intrathecal Drug Delivery
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1656
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Palsy; Multiple Sclerosis; Traumatic Brain Injury; Spinal Cord Injury
Keywords: Feasibility; SynchroMed II; Intrathecal catheter; Baclofen
MeSH Terms: conditions — Cerebral Palsy; Multiple Sclerosis; Brain Injuries, Traumatic; Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to record signatures from the fluid surrounding the spinal cord from people who have an implanted drug infusion system.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to record cerebrospinal fluid (CSF) signatures from subjects who have an implanted drug infusion system and who undergo clinical tests designed to troubleshoot possible catheter-related problems as part of their normal standard of care. Signatures will be correlated with physician-determined catheter status.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 12 years of age
* Have an implanted Medtronic drug infusion system for chronic intrathecal administration of drugs
* Report decreased therapeutic benefit, or show visible signs and/or symptoms of decreased therapeutic benefit
* Agree to undergo clinical tests designed to troubleshoot catheter-related problems or failure as a part of their normal standard of care
* Agree to provide signed informed consent.

Exclusion Criteria:

* Are currently enrolled or plan to enroll in another investigational drug or device trial
* Have participated in an investigational drug or device study within 30 days of the in-clinic visit
* Whose health status would, in the opinion of the Clinical Investigator, be jeopardized by participation in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with implanted Medtronic drug infusion system for chronic intrathecal administration, and who report decreased therepeutic benefit or who present with visible signs and/or symptoms of decreased therapeutic benefit, suggesting possible catheter-related problems.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Turner, MD, Principal Investigator — Goodman Campbell Brain and Spine; Michael Saulino, MD, Principal Investigator — Moss Rehab
Locations (2):
- United States (2):
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Moss Rehab, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Coffey RJ, Miesel K, Billstrom T. Cerebrospinal fluid pressure measurement in the ovine intrathecal space: a preliminary study towards the diagnosis of intrathecal drug administration catheter dislodgement or occlusion. Stereotact Funct Neurosurg. 2010;88(6):337-44. doi: 10.1159/000319034. Epub 2010 Aug 21. PMID 20733347
- [Result] Saulino M, Miesel K, Turner M, Cochran F, Stromberg K, Fehrmann E, Markert M. Can CSF pressure signals distinguish catheter complications from normal catheter function in subjects who experience loss of intrathecal baclofen therapy? Abstract submitted to the 11th World Congress of the International Neuromodulation Society (June 2013; Berlin).
- [Result] Saulino M, Turner M, Miesel K, Cochran FR, Stromberg K, Fehrmann E, Markert M, Spencer R. Can Cerebrospinal Fluid Pressure Detect Catheter Complications in Patients Who Experience Loss of Effectiveness With Intrathecal Baclofen Therapy? Neuromodulation. 2017 Feb;20(2):187-197. doi: 10.1111/ner.12471. Epub 2016 Aug 1. PMID 27477589

RESULTS

PARTICIPANT FLOW:
Groups:
- Intrathecal Pump Patients: Subjects previously implanted with an intrathecal pump who satisfied all inclusion and exclusion criteria, provided written informed consent, and had a needle inserted into the catheter access port of the implanted pump were considered to be enrolled in the study
Period: Overall Study
Arm/Group | Intrathecal Pump Patients
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intrathecal Pump Patients: Subjects who satisfied all inclusion and exclusion criteria, provided written informed consent, and had a needle inserted into the catheter access port of the implanted pump were considered to be enrolled in the study
Arm/Group | Intrathecal Pump Patients
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 37
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47
Infusion system spasticity treatment sub-indication [Number; unit: participants] — The primary treatment indication for all subjects was severe spasticity. This measure describes the treatment sub-indication for each subject.
  participants
    Cerebral palsy | 25
    Multiple sclerosis | 8
    Stroke | 3
    Brain injury | 3
    Spinal cord injury | 2
    Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Classification of Catheter Function by CSF Signatures vs. Physician's Standard Trouble-shooting Diagnosis
Description: Collect and characterize, by comparison with the physician's standard trouble-shooting diagnosis, CSF signatures recorded in subjects who have an infusion system who present with signs and/or symptoms of possible catheter-related problems or failure.
Time Frame: 1 day
Population: Subjects were excluded if the needle was not in the CAP, if they had a ventricular catheter, if the pressure sensor malfunctioned, or if there was an issue with the equipment
Measure: Number; unit: Subjects whose CSF data agree with MD Dx
Groups:
- Subjects With Normal Catheter Function by Physician Diagnosis: Subjects whose pressure data were analyzable and who received a trouble-shooting diagnosis of normal catheter function from the physician
- Subjects With Catheter Complications by Physician Diagnosis: Subjects whose pressure data were analyzable and who received a trouble-shooting diagnosis of catheter complication from the physician
Arm/Group | Subjects With Normal Catheter Function by Physician Diagnosis | Subjects With Catheter Complications by Physician Diagnosis
Number analyzed (Participants) | 19 | 18
Subjects whose CSF data agree with MD Dx | 13 | 16

2. Secondary Outcome: The Relationship Between Catheter Flow Resistance Check Data and Physician's Standard Trouble-shooting Diagnosis
Description: Characterize the relationship between pressure decay-to-baseline time (in seconds) and the physician's standard trouble-shooting diagnosis
Time Frame: 1 day
Population: Subjects were excluded if the needle was not in the CAP, if they had a ventricular catheter, if the pressure sensor malfunctioned, if there was an issue with the equipment, if the clamp was not open, or if the resistance check data were missing.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Subjects With Normal Catheter Function by Physician Diagnosis: Subjects whose catheter flow resistance check data were analyzable and who received a trouble-shooting diagnosis of normal catheter function from the physician
- Subjects With Catheter Complications by Physician Diagnosis: Subjects whose catheter flow resistance check data were analyzable and who received a trouble-shooting diagnosis of catheter complication from the physician
Arm/Group | Subjects With Normal Catheter Function by Physician Diagnosis | Subjects With Catheter Complications by Physician Diagnosis
Number analyzed (Participants) | 19 | 16
seconds | 6.4 (15.3) | 19.9 (18.1)

3. Secondary Outcome: The Relationship Between CSF Pressure Data and Physician's Standard Trouble-shooting Diagnosis During Physical Task Protocol: Cough
Description: Collect and characterize, by comparison with the physician's standard trouble-shooting diagnosis, the mean change in CSF pressure data during the physical task of a cough
Time Frame: 1 day
Population: Subjects were excluded if the needle was not in the CAP, if they had a ventricular catheter, if the pressure sensor malfunctioned, if there was an issue with the equipment, or if the subject was unable to cough.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Subjects With Normal Catheter Function by Physician Diagnosis: Subjects whose pressure data in response to cough were analyzable and who received a diagnosis of normal catheter function from the physician
- Subjects With Catheter Complications by Physician Diagnosis: Subjects whose pressure data in response to cough were analyzable and who received a diagnosis of catheter complication from the physician
Arm/Group | Subjects With Normal Catheter Function by Physician Diagnosis | Subjects With Catheter Complications by Physician Diagnosis
Number analyzed (Participants) | 18 | 17
mmHg | 21.0 (13.8) | 6.6 (6.7)

4. Secondary Outcome: The Relationship Between CSF Pressure Data and Physician's Standard Trouble-shooting Diagnosis During Physical Task Protocol: Valsalva
Description: Collect and characterize, by comparison with the physician's standard trouble-shooting diagnosis, the mean change in CSF pressure data during the physical task of a valsalva maneuver
Time Frame: 1 day
Population: Subjects were excluded if the needle was not in the CAP, if they had a ventricular catheter, if the pressure sensor malfunctioned, if there was an issue with the equipment, if the subject was unable to perform the valsalva, or if data were missing.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Subjects With Normal Catheter Function by Physician Diagnosis: Subjects whose pressure data in response to valsalva were analyzable and who received a diagnosis of normal catheter function from the physician
- Subjects With Catheter Complications by Physician Diagnosis: Subjects whose pressure data in response to valsalva were analyzable and who received a diagnosis of catheter complication from the physician
Arm/Group | Subjects With Normal Catheter Function by Physician Diagnosis | Subjects With Catheter Complications by Physician Diagnosis
Number analyzed (Participants) | 18 | 16
mmHg | 18.7 (12.8) | 4.8 (5.8)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout this research study, from time of subject enrollment to subject discontinuation. The minimum duration of subject follow-up was 47 days; the maximum was 287 days.
Description: All adverse events were collected for the duration of the study. No adverse events were associated with the measurement of CSF pressure energy, including insertion of the needle into the CAP and subsequent data acquisition lasting 6.3 ± 2.9 minutes (mean ± SD).
Arm/Group | Intrathecal Pump Patients
Serious Adverse Events (participants affected / at risk) | 14/47
Other Adverse Events (participants affected / at risk) | 6/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Pump Patients (N=47)
Implant site infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Muscle spasticity (Nervous system disorders) | 2 (2)
Nervous system disorder (Nervous system disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug withdrawal syndrom (General disorders) | 6 (7)
Implant site effusion (General disorders) | 1 (1)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Lumbar puncture headache (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Underdose (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intrathecal Pump Patients (N=47)
Incision site complication (General disorders) | 2 (2)
Muscle spasticity (Nervous system disorders) | 2 (3)
Wound dehiscence (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
"Normal" subjects who received intrathecal baclofen without experiencing catheter complications were not enrolled.

Subjects who received intrathecal drug delivery for chronic pain were not enrolled.

This was not a longitudinal study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days